CLINICAL TRIAL: NCT03238521
Title: Could the Intraoperative Radiation Exposure (Fluoroscopy) of Percutaneous Pedicle Screw Fixation be Reduced Using an Electronic Conductivity Device? A Prospective, Randomized Study
Brief Title: Could the Intraoperative Radiation Exposure (Fluoroscopy) of Percutaneous Pedicle Screw Fixation be Reduced Using an Electronic Conductivity Device?
Acronym: PEDI-PDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35RC16_9855_PEDI-PDS
Record Dates: First submitted 2017-07-25; First posted 2017-08-03 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classical pedicle finder (Active Comparator): Spinal osteosynthesis with classical pedicle finder
  Interventions: Procedure: Spinal osteosynthesis with classical pedicle finder
- pedicle finder with impedancemetry (Experimental): Spinal osteosynthesis with pedicle finder with impedancemetry
  Interventions: Procedure: Spinal osteosynthesis with pedicle finder with impedancemetry

INTERVENTIONS:
Procedure: Spinal osteosynthesis with classical pedicle finder — Posterior thoracic and lumbar osteosynthesis with classical pedicle finder
  Arms: classical pedicle finder
Procedure: Spinal osteosynthesis with pedicle finder with impedancemetry — Posterior thoracic and lumbar osteosynthesis with pedicle finder with impedancemetry
  Arms: pedicle finder with impedancemetry

SUMMARY:
To compare classical pedicle finder versus pedicle finder with impedancemetry on the perioperative radiation exposure of PPTLO. These two devices are already used in common practice.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 80 years-old;
* Patient with an indication of PPTLO for one or two segments
* Patient in a position to understand protocol information;
* Patient who received information about the protocol and who did not show opposition to participate

Exclusion Criteria:

* History of posterior spinal fusion surgery on the spinal level concerned by the study;
* Morbid obesity (body mass index greater than 35 kg / m²);
* Major incapable (safeguard of justice, guardianship) and persons deprived of liberty.
* Simultaneous participation in another research protocol involving the human person

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-11-11 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Dose area product in cGy.cm2 (DAP) | Surgery Day
  Dose area product in cGy.cm2 (DAP)

SECONDARY OUTCOMES:
Radiation duration in seconds (measured on the fluoroscope); | Surgery Day
  Radiation duration in seconds (measured on the fluoroscope);
Radiation rate | Surgery Day
  Radiation rate on:1 ring carried by the surgeon (passive dosimeter),1 passive dosimeter worn at the surgeon's eye level, 1 passive dosimeter on the fluoroscope,1 active dosimeter placed on the bust of the surgeon under the lead apron
Path of pedicle screws extracted from fluoroscopic images | Day 2 after surgery
  Trajectory of pedicle screws;
Operating time in minutes. | Surgery Day
  Operating time in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan LEBHAR, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Orthopedic surgery division, Rennes, France